CLINICAL TRIAL: NCT03573726
Title: Use of a Diurnal Indwelling Urethral Catheter to Improve Quality of Life for Patients With Spina Bifida and Spinal Cord Injury
Brief Title: Use of a Diurnal Indwelling Urethral Catheter to Improve Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Eric A Kurzrock, Professor of Urology and Pediatrics, Shriners Hospitals for Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 429063
Record Dates: First submitted 2018-05-08; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Spina Bifida; Neurogenic Bladder
MeSH Terms: conditions — Spinal Dysraphism; Urinary Bladder, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Technically N/A, Crossover Design (Other): Each participant underwent an evaluation during standard of care CIC use vs evaluations during use of the study intervention (CDIC).
  Interventions: Other: Closed diurnal indwelling catheter (CDIC)

INTERVENTIONS:
Other: Closed diurnal indwelling catheter (CDIC) — Each participant underwent an evaluation during standard of care CIC use vs evaluations during use of the study intervention (CDIC).

SUMMARY:
This is an interventional study examining the effects of closed diurnal indwelling catheterization (CDIC) for neurogenic bladder management.

DETAILED DESCRIPTION:
This is an interventional study examining the effects of indwelling diurnal catheter use in 10 to 21 year old individuals with neurogenic bladder due to Spina Bifida or spinal cord injury.Subject participation is expected to last up to 6 months.Eligible, interested patients will complete a pre-study visit for a clinical assessment by a pediatric urologist, informed consent completion and education regarding the diurnal use of indwelling foley catheters. Each patient will be screened to ensure that they have completed standard studies of urologic function within the last six months including a serum chemistry panel, renal ultrasound, KUB, and urodynamic studies. Within four weeks prior to study onset, a UA and culture, pad weighing test and voiding diary will be completed. After initiation of diurnal catheter use, weekly screening calls and adverse event screening will be completed by the study coordinator with involvement of a pediatric urologist for evaluation and management as required for all screens with responses concerning for either symptomatic urinary tract infection or adverse event. There will be clinical assessments at SHCNC by the nurse practitioner or pediatric urologist at Week 4, 12 and 24 of participation (adverse event assessment, quality of life questionnaire completion, pad weight tests, voiding diary completion and UA/ culture). At the Week 12 and 24 visits, a renal ultrasound will be completed.

The option that the investigators propose is novel and is the use of an indwelling urethral catheter placed in the morning, remaining in place for 8 hours ('diurnal' indwelling catheter). Bladder drainage will occur on a scheduled basis during the school day or workday by the simple opening of the closed catheter. After eight hours, each evening, the indwelling catheter will be removed with resumption of CIC. This would be a convenient and practical solution that could simultaneously avoid many of the risks associated with long-term indwelling urethral catheter use, while still allowing for the improved independence, convenience and privacy desired by youth with spina bifida or spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10 to 21 years at study entry
2. Primary diagnosis of Spina Bifida or Spinal Cord Injury with neurogenic bladder and established patients of a pediatric urologist in the Shriners Hospitals for Children multidisciplinary spina bifida clinic.
3. History of compliance with a CIC regimen.
4. Ability to understand and the willingness to sign a written informed consent document on the part of both the subject and guardian. A signed assent will be required, on the part of the subject, for all youth aged 10 to 17 years at the onset of study participation. In these cases, a parent or legal guardian must additionally sign a provision of informed consent. For subjects 18 years of age and older at the onset of study participation, only the subject must sign a provision of informed consent and HIPAA compliant research authorization.

Exclusion Criteria:

1. Age less than10 years and greater than 21 years at study entry
2. Greater than 2 diagnosed UTIs within last 12 months or symptomatic UTI at trial onset (UTI defined as the presence or ≥104 cfu/ml of a single bacterial strain in the presence of identified symptoms including but not limited to fever, flank or abdominal pain, change in urinary pattern or dysuria). Potential screened subjects with a symptomatic UTI at time of screening may be included after treatment of the UTI, followed by verification of symptom resolution and a negative culture result.
3. History of bladder augmentation
4. History of prior urethral surgery
5. History of urinary tract calculi
6. Diagnosis of high volume vesicoureteral reflux (grade 3 to 5) or moderate to severe (grade 3-4) hydronephrosis on pre-study imaging within 6 months of trial onset.
7. Diagnosis on urodynamics of >40mmHg detrusor end fill pressure (consistent with a poorly compliant bladder) on pre-study urodynamics within 6 months of trial onset.
8. Diminished renal function (GFR <60, consistent with CKD III) on pre-study laboratory assessment within 4 weeks prior to study onset.
9. Lack of a 5th grade minimum reading/writing level by the subject (and parent or guardian providing informed consent of <18 years of age at time of study onset)
10. Demonstrated lack of compliance with follow-up, with >2 missed urologic appointments in past year and/or lack of compliance with clean intermittent catheterization.
11. Pregnant women (all female participants must have a negative pregnancy test within 4 weeks prior to study onset).
12. Prisoners, institutionalized individuals or wards of the state.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Trust SF-36 | at baseline, week 4,12, and 24
  Quality of Life is measured by questionnaire Medical Outcomes Trust SF-36. The physical component and mental component summary measures were selected from the SF-36 questionnaire. It measures change from baseline on CIC to week 4 of CDIC use in health related quality of life. We obtained the SF-36 site license from Quality Metric (Lincoln, RI) and are utilizing the proprietary software for all composite analyses.

SECONDARY OUTCOMES:
Urinary continence | at baseline, week 4,12, and 24
  Urinary specific quality of life will be assessed by the validated King's Health Questionnaire (KHQ). The King's Health Questionnaire (KHQ) consists of two portions, 21 questions total, which address general health and the impact of incontinence including limitations to roles, physical, emotional, social and personal domains, sleep disturbance and incontinence severity. Differences in component summary scores will be assessed at each endpoint weeks 4, 12, and 24 and compared to baseline scores as noted for the SF-36.
PedsQL | at baseline, week 4,12, and 24
  Pediatric quality of life will be assessed by the PedsQL (pediatric quality of life) 4.0 Generic Core Scales includes scales that assess child self-report and parent proxy-report of generic core health outcomes from the physical, emotional, social and school domains. Outcome endpoints and analyses are as described for the SF-36 and KHQ above and will evaluate each summary domain score at 4, 12 and 24 weeks on trial in comparison to baseline evaluation.